CLINICAL TRIAL: NCT06683807
Title: The Effect of Glass Particle Contamination From Bupivacaine Ampules on Postdural Puncture Headache After Spinal Anesthesia for Cesarean Section: A Randomized, Double-Blind, Placebo-Controlled Clinical Trial
Brief Title: Postdural Puncture Headache After Spinal Anesthesia for Cesarean Section
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Seham Mohamed Moeen Ibrahim, Princible investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SM112024
Record Dates: First submitted 2024-11-07; First posted 2024-11-12 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Headache
MeSH Terms: conditions — Headache

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group T0 (Placebo Comparator): Parturients will receive spinal anesthesia for elective cesarean delivery with injection of 25 μg fentanyl plus 12.5 mg of hyperbaric bupivacaine 0.5% (2.5 mL) immediately after opening the bupivacaine ampule and directly after immediate aspiration with an unfiltered 3 ml syringe
  Interventions: Drug: Hyperbaric bupivacaine 0.5% (2.5 mL) aspirated immediately after opening the bupivacaine ampule
- Group T5 (Active Comparator): Parturients will receive spinal anesthesia for elective cesarean delivery with injection of 25 μg fentanyl plus 12.5 mg of hyperbaric bupivacaine 0.5% (2.5 mL) directly after 5 min' delayed aspiration from opening of the bupivacaine ampule with an unfiltered 3 ml syringe to allow glass particles to settle onto the bottom of the ampule
  Interventions: Drug: Hyperbaric bupivacaine 0.5% (2.5 mL) aspirated 5 minutes delayed after opening the bupivacaine ampule

INTERVENTIONS:
Drug: Hyperbaric bupivacaine 0.5% (2.5 mL) aspirated immediately after opening the bupivacaine ampule — Parturients will receive spinal anesthesia for elective cesarean delivery with injection of 25 μg fentanyl plus 12.5 mg of hyperbaric bupivacaine 0.5% (2.5 mL) immediately after opening the bupivacaine ampule and directly after immediate aspiration with an unfiltered 3 ml syringe
  Arms: Group T0
Drug: Hyperbaric bupivacaine 0.5% (2.5 mL) aspirated 5 minutes delayed after opening the bupivacaine ampule — Parturients will receive spinal anesthesia for elective cesarean delivery with injection of 25 μg fentanyl plus 12.5 mg of hyperbaric bupivacaine 0.5% (2.5 mL) directly after 5 min' delayed aspiration from opening of the bupivacaine ampule with an unfiltered 3 ml syringe to allow glass particles to settle onto the bottom of the ampule
  Arms: Group T5

SUMMARY:
Post-dural puncture headache (PDPH) is a potential and debilitating complication of spinal anesthesia in pregnant patients undergoing caesarean sections (CS), with a reported incidence of 0.5%-2% .

DETAILED DESCRIPTION:
Various methods for the management of PDPH are present including proper hydration, maintaining a supine posture, caffeine, paracetamol, nonsteroid anti-inflammatory drugs (NSAID), theophylline, opioids like morphine and fentanyl, with the only clearly effective treatment being the epidural blood patch.

Glass particle contamination is known to occur on opening single-dose drug ampoules. Although supporting data are lacking, intrathecal drug administration during subarachnoid blocks and chemotherapy with glass particle contamination is potentially hazardous,

ELIGIBILITY:
Inclusion Criteria:

* Parturient with American Society of Anesthesiologists (ASA) class I or II
* Age: 20-45 years old
* A full-term pregnant female undergoing elective cesarean section under spinal anesthesia

Exclusion Criteria:

* Contraindications to regional anesthesia (coagulopathy, infection at the needle insertion site)
* History of Migraines or persistent headache
* Known hypersensitivity to local anesthetics
* Body mass index (BMI > 35 kg/m2)
* Hypertensive disorders of pregnancy
* Emergency cesarean section
* Cardiorespiratory, hepatic, or renal impairment
* History of a cerebrovascular accident, neurologic or psychological disorders
* Uncontrolled hypertension
* Spinal column surgery, chronic opioid consumption
* Patients with more than one single attempt and patients with blood loss over 1000 mL who will need additional fluid supplementation or blood transfusion
* Patient refusal

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 55 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
The incidence of post-dural puncture headache (PDPH) | The first 120 hours during the post-partum period.
  Assessed using the visual analog score of pain which ranges from 0-10, where 0 = no pain and 10 = maximum worst pain

CONTACTS AND LOCATIONS:
Overall Officials: Seham M Moeen, MD, Principal Investigator — Assiut University